CLINICAL TRIAL: NCT05882565
Title: A Brief Online Mindfulness Intervention for Indonesian Undergraduate Students: A Randomized Controlled Trial Protocol
Brief Title: A Brief Online Mindfulness Intervention: An RCT Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ka Yan (Other)
Collaborators: Radboud University, The Netherlands (Unknown)
Responsible Party: Sponsor-Investigator, Ka Yan, Lecturer at Universitas Kristen Maranatha, Maranatha Christian University
Organization: Maranatha Christian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7/KEP/II/2021
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Stress; Anxiety; Depression
Keywords: stress; anxiety; depression; mindfulness; repetitive negative thinking; undergraduate students; Indonesia
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfuness training group (Experimental): This is a group that will receive mindfulness intervention for 14 days. Participants in this group will also be asked baseline, daily and post questions, as well as follow up questions (3 months after the intervention). During the intervention, they can fill out an optional daily journal.
  Interventions: Behavioral: A brief (14-day) online mindfulness intervention
- Psychoeducation group (Active Comparator): This is a group that will receive psychoeducation intervention for 14 days. Participants in this group will also be asked baseline, daily and post questions, as well as follow up questions (3months after the intervention). During the intervention, they can fill out an optional daily journal.
  Interventions: Behavioral: Psychoeducation online
- Waitlist control group (No Intervention): This is a group that will not receive any training, however, this group will be asked several questions (baseline, daily and post questions, as well as follow up questions (3-months later)). They can also fill out an optional daily journal.

INTERVENTIONS:
Behavioral: A brief (14-day) online mindfulness intervention — The content of the online mindfulness intervention is based on studies by Cavanagh et al. (2013, 2018). There is an approximately 10-minute audio tutorial that participants will listen to daily for 14 days. In the first week, participants will be instructed to apply their learned mindfulness skills to their daily activities. In the second week, they will continue practicing by learning to walk in a mindful manner.
  Arms: Mindfuness training group
Behavioral: Psychoeducation online — The online psychoeducation was modified from the study by Harrer et al (2019, 2021).
  This intervention consists of 14 audio tutorials about stress for 14 days, each lasting approximately 10 minutes. Additionally, there is a text version of each audio tutorial, which can be accessed by participants after listening to the audio.
  Arms: Psychoeducation group

SUMMARY:
University students often experience emotional distress that originates from inside or outside academia, and for which treatment would be welcome. Research has shown that mindfulness can help people to reduce stress, anxiety and depression. Furthermore, a thinking style that focuses excessively on negative content (repetitive negative thinking; RNT) has consistently been found to be a mediator of the effects of mindfulness on decreasing stress, anxiety and depression. With this study, we want to 1) investigate the effects of mindfulness on stress, anxiety, depression, and RNT in Indonesian sample of undergraduate students and 2) investigate the mediating role of RNT.

DETAILED DESCRIPTION:
Time in university is a generally stressful period of life as a lot of students may face challenges both inside and outside academia. In Indonesia, the majority of undergraduate students (40-80%) reports severe to extremely severe levels of stress, anxiety and depression. Nevertheless, only few young people in Indonesia (< 5%) receive treatment due to the unavailability of mental healthcare facilities and high treatment costs. In addition, Indonesian students tend to not seek help from others when experiencing mental health problems, as sharing personal or family experiences about mental issues is generally perceived as embarrassing. A meta-analytic review concluded that online mindfulness has a large effect on reducing stress, and a small but significant beneficial impact on depression and anxiety. A recent systematic review showed that a brief online mindfulness intervention can offer positive mental health outcomes (i.e., reduction of stress, anxiety and depressive symptoms) for both clinical and non-clinical samples. Repetitive negative thinking (RNT), defined as a thinking style that focuses excessively on negative content, has consistently been found to be a mediator of the effects of mindfulness on stress reduction and the amelioration of anxiety and/or depressive symptoms. First, this study aims to investigate the effects of a brief (14-day) online mindfulness intervention on stress, anxiety, depressive symptoms and repetitive negative thinking (RNT) in an Indonesian sample of undergraduate students. It is hypothesized that participants in the mindfulness training and active control (psychoeducation) conditions will report less stress, anxiety, depressive symptoms and RNT after the intervention compared to the waitlist control condition. The psychoeducation intervention has the same structure and length as the mindfulness training, but the content differs as it does not involve skills training. Hence, psychoeducation can decrease mental health complaints, but, in line with previous studies, it is hypothesized that it will be less effective in reducing stress, anxiety and depressive symptoms than the mindfulness training. Second, this study aims to investigate the mediating role of RNT. That is, we study whether changes in RNT (i.e., a reduction) serve as a potential working mechanism through which mindfulness achieves its effect. It is hypothesized that RNT mediates the effects of mindfulness on stress, anxiety, and depressive symptoms.

ELIGIBILITY:
Inclusion criteria:

* Being admitted to one of the universities in Indonesia
* Having good eyesight and hearing
* Access to the internet and familiarity in navigating the internet

Exclusion criteria:

* Practicing yoga/ meditation/ mindfulness regularly
* Receiving psychological treatment at the time of study enrolment
* Current alcohol or drug abuse

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale-21 (DASS-21; Lovibond & Lovibond, 1995) | 2 weeks-3 months
  DASS-21will be administered to measure depressive symptoms, anxiety and stress. It consists of 21 items that have to be rated on a four-point Likert scale (0 = 'did not apply to me at all' to 4 = 'applied to me very much or most of the time'.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ: Baer et al., 2006) | 2 weeks-3 months
  Change in state mindfulness will be measured using The FFMQ. It includes 39 items, which have to be rated on five-point Likert scale (1 = 'never or very rarely true' to 5 = 'very often or always true'). It includes five components : observing, describing, nonjudging, non reactivity, and acting with awareness.
Perseverative Thinking Questionnaire (PTQ) | 2 weeks-3 months
  Changes in RNT will be measured using The PTQ. The questionnaire (Ehring et al., 2011) is distributed for the trait assessment of repetitive negative thinking, which includes 15-items rated on a five-point Likert scale (1 = 'never' to 5 = 'almost always').
Momentary repetitive negative thinking | 2 weeks (daily)
  There are five items to assess momentary repetitive negative thinking. These items inquire about thinking patterns related to feelings, problems, worries, recurring thoughts, and being stuck on certain issues. Each question should be answered using a seven-point Likert scale, with responses ranging from 1 = 'never' to 7 = 'every time'.
Mood questions | 2 weeks (daily)
  To be able to check training adherence and training performance, questions regarding context (i.e., (1) Are you in a quiet room at the moment, (2) Are you sitting in a comfortable position with your feet flat on the floor [for mindfulness training condition only] and company (i.e., (3) Are you surrounded by company?) will be asked. These questions can be answered with a 'yes' or 'no'.
Daily Journal | 2 weeks (daily)
  In order to obtain additional information about participants' experiences, thoughts, feelings or difficulty regarding the intervention, we will ask them to fill out an (optional) daily journal. Participants can write in the journal at the end of the (everyday) training.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Spijker, Professor, Principal Investigator — Radboud University, Propersona Institute for Integrated Mental Health Care; Ka Yan, Master, Study Chair — Universitas Kristen Maranatha-Indonesia, Radboud University-The Netherlands; Cilia Witteman, Professor, Study Chair — Radboud University, The Netherlands; Nessa Ikani, Doctor, Study Chair — Radboud University, Pro Persona, Tilburg University-The Netherlands; Cleoputri Yusainy, Study Chair — Brawijaya University-Indonesia
Locations (1):
- Universitas Kristen Maranatha, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: 6 months after publication of the manuscript

REFERENCES:
- [Derived] Yan K, Ikani N, Yusainy C, Witteman C, Spijker J. A brief online mindfulness intervention: study protocol for Indonesian undergraduate students, a randomized controlled trial. Trials. 2025 May 13;26(1):155. doi: 10.1186/s13063-025-08858-y. PMID 40361160